CLINICAL TRIAL: NCT00049790
Title: Safety and Efficacy Study of rhAngiostatin Administered in Combination With Paclitaxel and Carboplatin to Patients With Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Purpose: Treatment
Other Study IDs: ANG-CL-004
Record Dates: First submitted 2002-11-13; First posted 2002-11-15 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Advanced non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Carboplatin

INTERVENTIONS:
Drug: recombinant human Angiostatin protein
Drug: paclitaxel
Drug: carboplatin

SUMMARY:
The purpose of this study is to determine the safety and efficacy of rhAngiostatin protein administered in combination with paclitaxel and carboplatin to patients with non-small-cell lung cancer.

ELIGIBILITY:
Inclusion:

* Histological or cytological confirmed Stage IIIB NSCLC with malignant pleural effusions, or Stage IV NSCLC or recurrent NSCLC
* No previous chemotherapy for NSCLC
* Have one lesion that is bidimensionally measurable by physical exam, MRI, or CT greater than 1 cm in diameter
* Specified lab parameters
* Life expectancy of at least 12 weeks
* ECOG performance status of 0 or 1
* Understand requirements of study
* Agree to use effective contraceptive methods

Exclusion:

* Have CNS metastases
* Have any active cancer in addition ot NSCLC
* Participated in clinical trial involving conventional or investigational drugs within previous 4 weeks
* Have any contraindication to paclitaxel or carboplatin
* Have had Grade 3 or greater peripheral neuropathies
* Be pregnant or lactating
* Have a history of myocardial infarction or angina pectoris/angina in the last 6 months
* Have had significant (30 mL or more) hemoptysis with the past 3 months
* Have an active infection
* Have a history of bleeding diathesis, hypercoagulable condition, or an active bleeding disorder
* Be receiving concurrent treatment with therapeutic doses of heparin or coumadin
* Have had major surgery within 4 weeks of stating therapy
* Have additional uncontrolled serious medical conditions or psychiatric illness
* Received rhAngiostatin in other clinical protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2004-12

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana Cancer Pavilion, Indiana University, Indianapolis, Indiana, United States